CLINICAL TRIAL: NCT05985031
Title: Does Reciprocal Inhibition, a Rehabilitation Technique, Convert to Reciprocal Facilitation in Patients With Upper Motor Neuron Lesions?
Brief Title: Reciprocal Inhibition Versus Reciprocal Facilitation In Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Kökçe, assistant doctor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RIVRFSCIP
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord; motor neuron; Spasticity
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity | interventions — H-Reflex

STUDY DESIGN:
Intervention Model Description: Group I. Spinal cord injuries Group II. Healthy Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal cord injuries (Experimental): This was the patient group. Achilles tendon hits were performed for eliciting the soleus T reflex while the ankle was in neutral, dorsiflexion, and plantar flexion. Surface and multi-unit EMG recordings were taken from the anterior and soles muscles of the tibialis during the tendon tapping.
  Interventions: Diagnostic Test: Tendon tap; Diagnostic Test: Tibial nerve stimulation
- Healthy Control (Active Comparator): This was the healthy control group. Achilles tendon hits were performed for eliciting the soleus T reflex while the ankle was in neutral, dorsiflexion, and plantar flexion. Surface and multi-unit EMG recordings were taken from the anterior and soles muscles of the tibialis during the tendon tapping.
  Interventions: Diagnostic Test: Tendon tap; Diagnostic Test: Tibial nerve stimulation

INTERVENTIONS:
Diagnostic Test: Tendon tap — While examining the T reflex, the ankle was held passively in neutral, dorsiflexion and plantar flexion positions by the investigator.
  Other Names: T-reflex
Diagnostic Test: Tibial nerve stimulation — H-reflex responses were examined by tibial nerve stimulation
  Other Names: H-reflex

SUMMARY:
Reciprocal inhibition is a medulla spinalis control mechanism that facilitates motor activities in healthy people. As the agonist muscle contracts, the antagonist muscle is inhibited so that the agonist action can take place properly. In the literature, there are studies showing that in patients with upper motor neuron lesions, this reverses, and reciprocal facilitation occurs instead of inhibition. However, there is no clear situation in this regard, there is a need for more methodologically sound studies. Our aim in this study is to investigate the presence of reciprocal facilitation in patients with spinal cord lesions (SCL).

DETAILED DESCRIPTION:
Reciprocal inhibition is a spinal segmental control mechanism that facilitates motor activities in healthy people and is also used in treating spasticity. Considering the current literature, there are some studies claiming that this is reversed in patients with upper motor neuron lesions and that there is reciprocal facilitation instead of inhibition. However, the proposed evidence is not convincing. Our aim in this study was to investigate the presence of reciprocal facilitation in detail in patients with upper motor neuron lesions. This study was conducted in five patients with spinal cord lesions and five healthy individuals. Both the tibialis anterior and soleus muscles of the cases were recorded using surface and multi-motor unit electromyography (EMG) electrodes. To elicit an H reflex in the soleus muscle, an electric current was delivered through the popliteal fossa using the monopolar technique. The Achilles tendon was tapped with the reflex hammer to elicit a T reflex. Since the H-reflex and T-reflex responses were detected in the tibialis anterior muscle surface and multi-motor unit EMG recordings, the findings were evaluated as direct stimulation, cross-talk, and reciprocal facilitation. Methodologically, This research aimed to be a guiding study for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spinal cord injury between the ages of 18-60
* A minimum of 6 months of SCL history
* Soleus spasticity

Exclusion Criteria:

* Patients with premorbid neuromuscular disease
* History of autonomic dysreflexia
* Patients in the spinal shock period
* Those who have a coronavirus disease clinic
* Less than 2 hours sitting tolerance

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Reciprocal Inhibition | up to 2 weeks
  H reflex and T reflex tests were performed in the soleus and tibialis anterior muscle, and it was evaluated whether there was reciprocal inhibition in the tibialis anterior muscle.

SECONDARY OUTCOMES:
H-reflex | up to 2 weeks
  Electric current was delivered through the popliteal fossa to tibial nerve for eliciting the soleus H-reflex
T-reflex | up to 2 weeks
  The Achilles tendon was hit with using a reflex hammer to elicit the soleus T-reflex.

CONTACTS AND LOCATIONS:
Overall Officials: İLHAN KARACAN, MD, Prof, Study Director — İstanbul Physical Therapy Rehabilitation Training & Research Hosptial
Locations (1):
- İstanbul Physical Therapy Training and Research Hospital, Istanbul, Turkey (Türkiye)